CLINICAL TRIAL: NCT01250847
Title: Phase IV Study of Effects of 'Seroquel-XR' on the Improvement of Neurocognitive Function in People At-risk Mental States(ARMS)
Brief Title: Effects of 'Seroquel-XR' on the Improvement of Neurocognitive Function in People At-risk Mental States(ARMS)
Acronym: ES-ARMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Suk Kyoon An, Severance Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARMS-4001
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2010-11

CONDITIONS: Abnormal Mental State; Schizophrenia
Keywords: ARMS; Ultra High Risk; Quetiapine; Verbal memory
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Seroquel-XR (Experimental): The subjects At-Risk Mental States will be treated with Quetiapine(Seroquel-XR) from baseline to end of trial.
  Interventions: Drug: Quetiapine(Seroquel-XR) 50~800mg a day
- Schizophrenia Comparator (Experimental): The subject with schizophrenia will be treated with standard treatment
  Interventions: Drug: Quetiapine(Seroquel-XR) 50~800mg a day
- Healthy Control Comparator (No Intervention): The subjects will not be required to treat
  Interventions: Drug: Quetiapine(Seroquel-XR) 50~800mg a day

INTERVENTIONS:
Drug: Quetiapine(Seroquel-XR) 50~800mg a day — The only ARMS subjects will be given 50~800mg Seroquel-XR once daily for total of 12 weeks.
  Other Names: Quetiapine(Seroquel-XR)

SUMMARY:
The primary objective of this study is to assess the effects of 'Seroquel-XR' on the verbal learning ability in people with at-risk mental state (ARMS) over a 12 week period. The verbal learning ability will be indexed by delayed free recall score of CVLT(California Verbal learning Test), a standard neuropsychological verbal memory tests.

The secondary objective is to assess the effects of 'Seroquel-XR' on other cognitive function and psychiatric symptoms including psychotic, anhedonic symptoms, and impulsivity. The cognitive function abilities will be measured by standard neuropsychological tests as follows;

* Working memory: verbal & spatial 2-back test
* Attention: Digit Span, 3-7 CPT(Continuous Performance Test)
* Executive function: WCST (Wisconsin Card Sorting Test)
* Visuo-spatial ability: Rey Complex Figure Task copy
* Visuomotor speed and planning: Trail making test A & B
* Verbal fluency: Controlled Oral Word Association Test(COWAT) The scales of psychiatric symptoms which will be used are as follows;
* Psychotic symptoms: Scales of Prodromal scales (SOPS), Positive and negative syndrome scale (PANSS)
* Anhedonia: Social Anhedonia Scale (SAS), Physical Anhedonia Scale (PAS)
* Social cognition: Ambiguous Intention Hostility Questionnaire (AIHQ)
* Impulsivity: Barrett Impulsivity Scale (BIS)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Male and female aged 20 to 35 years
3. Able to understand and comply with the requirements of the study

   ARMS:
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
5. ARMS was diagnosed by Structured Interview for Prodromal Syndrome (SIPS) .

Schizophrenia subjects:

4. Schizophrenia was diagnosed by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV). Patients with schizophrenia had to have been ill no more than 5 years. Subjects had to be clinically stable and on stable antipsychotic therapy for at least 4 weeks prior to baseline study.

Normal control:

4. Healthy volunteers who had no history of psychiatric illness and had no first degree relative with psychotic symptoms were included for normal controls.

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria. However, in the case of ARMS, psychotic disorder NOS, major depressive disorder, obsessive-compulsive disorder, and social phobia would be allowed.
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
12. Involvement in the planning and conduct of the study
13. Previous enrolment or randomisation of treatment in the present study.
14. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
15. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) more than 8.5 percent.

    Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.

    Not under physician care for DM Physician responsible for patient's DM care has not indicated that patient's DM is controlled.

    Physician responsible for patient's DM care has not approved patient's participation in the study Has not been on the same dose of oral hypoglycaemic drug(s) and(or) diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.

    Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10 percent above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
16. An absolute neutrophil count (ANC) of 1.5 folded 109 per liter

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
California Verbal Learning Test | Baseline
  Change from baseline in Verbal learning ability measured by CVLT at 12 weeks
California Verbal Learning Test | 12th week
  Change from baseline in Verbal learning ability measured by CVLT at 12 weeks

SECONDARY OUTCOMES:
verbal & spatial 2-back test, Digit Span, 3-7 CPT, WCST, Rey-CFT, TMT A & B, COWAT, SOPS, PANSS, SAS, PAS, AIHQ, BIS | Baseline
  Change from baseline in Working Memory etc. at 12 weeks
verbal & spatial 2-back test, Digit Span, 3-7 CPT, WCST, Rey-CFT, TMT A & B, COWAT, SOPS, PANSS, SAS, PAS, AIHQ, BIS | 12th week
  Change from baseline in working memory etc. at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suk Kyoon An, MD, Ph D, Principal Investigator — Severance Hospital
Locations (2):
- South Korea (2):
  - Severance Mental Health Hospital, Gwangju
  - Severance Hospital, Seoul